CLINICAL TRIAL: NCT00225511
Title: Phase III Multi-Center, Double-Blind, Comparative Study of Effexor XR for the Treatment of Depression
Brief Title: Study Evaluating Effexor XR for Major Depression.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0600B1-816
Record Dates: First submitted 2005-09-12; First posted 2005-09-23 (Estimated); Last update posted 2007-05-24 (Estimated); Status verified 2007-05

CONDITIONS: Depression
Keywords: Depression
MeSH Terms: conditions — Depression | interventions — Venlafaxine Hydrochloride; Milnacipran

INTERVENTIONS:
Drug: Effexor XR
Drug: Milnacipran

SUMMARY:
Study Evaluating Effexor XR for Major Depression.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with major depression based on DSM-IV-TR
* Patients having minimal total score of 18 on the HAM-D17 and minimal score of 2 on the item of "depressed mood" at the baseline.

Exclusion Criteria:

* Patients with schizophrenia or any other psychotic disorder
* Patients with history or presence of bipolar disorder

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 590 (Estimated)
Dates: Start 2004-06

PRIMARY OUTCOMES:
Response rate of HAM-D17 (Hamilton Rating Scale for Depression) at the final-on-therapy.

SECONDARY OUTCOMES:
Difference of total score of HAM-D17 between baseline and final-on-therapy.
Remission rate of HAM-D17 at the final-on-therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (43):
- Japan (43):
  - Nagoya, Aichi-ken
  - Ichikawa, Chiba
  - Fukuoka, Fukuoka
  - Kasuga, Fukuoka
  - Kitakyushu, Fukuoka
  - Kurume, Fukuoka
  - Ohnojyo, Fukuoka
  - Hiroshima, Hiroshima
  - Kure, Hiroshima
  - Otaru, Hokkaido
  - Sapporo, Hokkaido
  - Nishinomiya, Hyōgo
  - Tsuchiura, Ibaragi
  - Tsukuba, Ibaragi
  - Kanazawa, Ishikawa-ken
  - Hanamaki, Iwate
  - Kawasaki, Kanagawa
  - Sagamihara, Kanagawa
  - Yokohama, Kanagawa
  - Kikuchi, Kumamoto
  - Nagasaki, Nagasaki
  - Ohmura, Nagasaki
  - Kashihara, Nara
  - Jyo-etsu, Niigata
  - Beppu, Ohita
  - Moriguchi, Osaka
  - Osaka, Osaka
  - Sayama, Osaka
  - Saitama, Saitama
  - Hamamatsu, Shizuoka
  - Adachi-ku, Tokyo
  - Bunkyo-ku, Tokyo
  - Chiyoda-ku, Tokyo
  - Itabashi-ku, Tokyo
  - Kodaira, Tokyo
  - Meguro-ku, Tokyo
  - Minato-ku, Tokyo
  - Nakano-ku, Tokyo
  - Ohta-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Shinjuku, Tokyo
  - Tachikawa, Tokyo
  - Toshima-ku, Tokyo